CLINICAL TRIAL: NCT02293655
Title: The Effects of ADHD Medication (TEAM) Study: Neurobehavioral Effects of Abrupt Methylphenidate Discontinuation
Brief Title: The Effects of ADHD Medication (TEAM) Study
Acronym: TEAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADHDMedTEAMStudy
Record Dates: First submitted 2014-10-29; First posted 2014-11-18 (Estimated); Results first posted 2022-02-04 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-11

CONDITIONS: ADHD
Keywords: ADHD; inattention; hyperactivity; methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MPH Discontinuation (Placebo Comparator): 1. Double-blind (DB) placebo-controlled 4-week methylphenidate (MPH) titration trial. Pts will receive 3 active dosages of MPH (children <25kg: 18mg, 27mg, 36mg; children >25kg: 18mg, 36mg, 54mg for) as well as 1 random week of placebo, given qAM. Pts will begin on the lowest dose (or a randomized placebo week) and proceed through all dose conditions in an incremental fashion.
  2. DB 4-week MPH maintenance phase. The clinician, parent, and teacher ratings of behavior and side effects from the titration trial weeks will be graphed. Two doctors will blindly review the graphs and judge which week was the optimal dose week. Pts will then receive their optimal dose of MPH (qAM) for 4 weeks.
  3. DB 4-week MPH Discontinuation Phase. Pts in this arm will receive placebo (qAM).
  Interventions: Drug: OROS-Methylphenidate (MPH)
- Sustained MPH (Active Comparator): 1. Double-blind (DB) placebo-controlled 4-week methylphenidate (MPH) titration trial. Pts will receive 3 active dosages of MPH (children <25kg: 18mg, 27mg, 36mg; children >25kg: 18mg, 36mg, 54mg for) as well as 1 random week of placebo, given qAM. Pts will begin on the lowest dose (or a randomized placebo week) and proceed through all dose conditions in an incremental fashion.
  2. DB 4-week MPH maintenance phase. The clinician, parent, and teacher ratings of behavior and side effects from the titration trial weeks will be graphed. Two doctors will blindly review the graphs and judge which week was the optimal dose week. Pts will then receive their optimal dose of MPH (qAM) for 4 weeks.
  3. DB 4-week MPH Discontinuation Phase. Pts in this arm will continue their optimal MPH dose (qAM).
  Interventions: Drug: OROS-Methylphenidate (MPH)

INTERVENTIONS:
Drug: OROS-Methylphenidate (MPH) — OROS-methylphenidate will be taken orally once daily at doses that have been approved for the study age group by the U.S. FDA.
  Other Names: Concerta

SUMMARY:
This study evaluates the effects of receiving and then discontinuing methylphenidate (MPH) in children with ADHD. After receiving MPH for 8 weeks, participants will be randomized to either discontinue MPH (and receive placebo) OR remain on MPH for 4 weeks.

DETAILED DESCRIPTION:
The stimulant methylphenidate (MPH) is the most commonly prescribed psychoactive medication in children. An abundance of studies attest to the efficacy of MPH for attenuating inattentive, hyperactive, and impulsive symptoms in children with ADHD. Despite its efficacy, most children with ADHD who are prescribed MPH have poor continuity of treatment for a variety of reasons, including forgetting to administer the medication and delays obtaining refills. In addition, it is an accepted clinical practice for physicians to omit MPH for periods of time, such as during the summer or on weekends (i.e., drug holidays). Since MPH discontinuation is considered to be benign, many clinicians do not employ any special procedures or inform families of any special precautions in regard to its cessation. However, increasing evidence suggests that the pharmacological effects of MPH cause lasting changes in brain neurochemistry that persist beyond medication discontinuation. Moreover, these neurobiological effects of discontinuation appear to have neurobehavioral consequences. There is a critical need to better understand the breadth and magnitude of the neurobehavioral effects caused by MPH discontinuation as well as to better understand the temporal trajectory of these deleterious effects. Hence, the primary goal of the proposed research is to conduct the first randomized, double-blind, placebo-controlled trial specifically designed to study the negative effects of MPH discontinuation at multiple time points. 180 children diagnosed with ADHD will participate across two recruitment sites. After undergoing a 4-week MPH titration trial and 4-week MPH maintenance phase, participants will be randomized to either discontinue MPH (and receive placebo) OR remain on MPH for 4 weeks. Comprehensive multi-time point, multi-informant (parents, teachers, study staff) and multi-modal (behavior/mood/affect ratings scales, direct behavior observations, standardized testing) assessments will be used to assess a broad range of neurobehavioral outcomes. We will examine the magnitude and time course of effects of MPH discontinuation on behavioral as well as cognitive and academic functioning in children with ADHD. Furthermore, we will examine moderators of the adverse effects of MPH discontinuation on these outcomes to aid in the identification of those who are at increased risk.

ELIGIBILITY:
Inclusion Criteria:

1. ADHD Diagnostic Status: Meets DSM-V criteria for ADHD, with Clinical Global Impression (CGI) rating corresponding to at least "moderately ill."
2. Cognitive and Academic Functioning: Intelligence Quotient (IQ) of >80 as estimated by Vocabulary and Block Design subtests of the Wechsler Intelligence Scale for Children-4th Edition and scaled scores >80 on the Wechsler Individual Achievement Test-2nd edition Reading and Math subtests
3. Physical Health: Physical exam and ECG findings are judged to be normal for age and sex by study physician and/or medical consultant, and there is no co-existing condition for which MPH is contraindicated 4. School: Enrolled in a school setting rather than a home-school program. This ensures that we can obtain parent and teacher ratings from separate individuals for diagnosis and outcome assessment

Exclusion Criteria:

1. Psychiatric Medications: Current or prior use of any medication for psychological/psychiatric problems
2. Behavioral Interventions: Current active participation in ADHD-related behavioral interventions, given that improvements due to these interventions may confound our group comparisons
3. Psychiatric or Neurobehavioral Conditions: Children with mania/hypomania, schizophrenia, or severe depressive disorder, as determined by the K-SADS, will be excluded since ADHD medications may not be an appropriate first line of treatment for children with these comorbid disorders
4. Organic Brain Injury: History of head trauma, neurological disorder (including epilepsy), or other disorder affecting brain function due to potential differences in neurophysiology of ADHD phenotype
5. Cardiovascular Risk Factors: Children with a personal history or family history of cardiovascular risk factors will be excluded, or given the option of participating in the study after obtaining an EKG and verification from a pediatric cardiologist regarding the safety of their participation in a trial of methylphenidate. In this case, families will be responsible for the costs of EKG and any necessary cardiologist evaluation
6. Pregnancy: The safety of MPH use during pregnancy has not been established

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 204 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya E. Froehlich, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Seattle Children's Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The number Enrolled (those who signed informed consent) differs from the number who Started in the Participant Flow module because: 1) some children who signed informed consent were determined to be ineligible after having formal assessment for study inclusion, 2) some children were unable to learn to swallow the study pill so could not start protocol participation, 3) some families changed their minds about participating after signing informed consent but before starting study procedures.
Groups:
- MPH Discontinuation: 1. Double-blind (DB) placebo-controlled 4-week methylphenidate (MPH) titration trial. Pts will receive 3 active dosages of MPH (children <25kg: 18mg, 27mg, 36mg; children >25kg: 18mg, 36mg, 54mg for) as well as 1 random week of placebo, given qAM. Pts will begin on the lowest dose (or a randomized placebo week) and proceed through all dose conditions in an incremental fashion.
  2. DB 4-week MPH maintenance phase. The clinician, parent, and teacher ratings of behavior and side effects from the titration trial weeks will be graphed. Two doctors will blindly review the graphs and judge which week was the optimal dose week. Pts will then receive their optimal dose of MPH (qAM) for 4 weeks.
  3. DB 4-week MPH Discontinuation Phase. Pts in this arm will receive placebo (qAM).
  OROS-Methylphenidate (MPH): OROS-methylphenidate will be taken orally once daily at doses that have been approved for the study age group by the U.S. FDA.
- Sustained MPH: 1. Double-blind (DB) placebo-controlled 4-week methylphenidate (MPH) titration trial. Pts will receive 3 active dosages of MPH (children <25kg: 18mg, 27mg, 36mg; children >25kg: 18mg, 36mg, 54mg for) as well as 1 random week of placebo, given qAM. Pts will begin on the lowest dose (or a randomized placebo week) and proceed through all dose conditions in an incremental fashion.
  2. DB 4-week MPH maintenance phase. The clinician, parent, and teacher ratings of behavior and side effects from the titration trial weeks will be graphed. Two doctors will blindly review the graphs and judge which week was the optimal dose week. Pts will then receive their optimal dose of MPH (qAM) for 4 weeks.
  3. DB 4-week MPH Discontinuation Phase. Pts in this arm will continue their optimal MPH dose (qAM).
  OROS-Methylphenidate (MPH): OROS-methylphenidate will be taken orally once daily at doses that have been approved for the study age group by the U.S. FDA.
Period: Overall Study
Arm/Group | MPH Discontinuation | Sustained MPH
Started | 92 | 17
Completed | 85 | 15
Not Completed | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MPH Discontinuation | Sustained MPH | Total
Number analyzed (Participants) | 92 | 17 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 92 | 17 | 109
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 6 | 37
  Male | 61 | 11 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 1 | 9
  Not Hispanic or Latino | 84 | 16 | 100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 73 | 15 | 88
  More than one race | 10 | 0 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 92 | 17 | 109
Parent Vanderbilt ADHD Total Symptom Score [Mean (Standard Deviation); unit: score on a scale] — Parent Vanderbilt ADHD Rating Scale Total Symptom Score: minimum=0, maximum=54, higher scores indicate more/worse symptoms
  score on a scale | 36.2 (8.3) | 34.6 (10.9) | 36.0 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Parent ADHD Total Symptom Scores
Description: Parent Vanderbilt ADHD Rating Scale Total Symptom Score, minimum=0, maximum=54, higher scores indicate more/worse ADHD symptoms
Time Frame: baseline, study weeks 8, 9, 10, 12
Population: There was some attrition and missing data at different data collection points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MPH Discontinuation | Sustained MPH
Number analyzed (Participants) | 92 | 17
score on a scale
  Baseline | 36.2 (8.3) | 34.6 (10.9)
  Maintenance Visit (week 8): number analyzed (Participants) | 87 | 15
  Maintenance Visit (week 8) | 17.6 (8.8) | 15.3 (8.3)
  Randomization 1 (week 9): number analyzed (Participants) | 65 | 9
  Randomization 1 (week 9) | 16.5 (12.0) | 12.3 (10.4)
  Randomization 2 (week 10): number analyzed (Participants) | 82 | 15
  Randomization 2 (week 10) | 23.8 (11.6) | 14.3 (8.3)
  Randomization 3 (week 12): number analyzed (Participants) | 82 | 15
  Randomization 3 (week 12) | 25.2 (11.6) | 17.3 (12.3)
Statistical Analysis 1: Comparison: MPH Discontinuation vs Sustained MPH; Compared at Baseline Time point; Test type: Superiority; p = 0.55, t-test, 2 sided; Mean Difference (Final Values) = 1.6, Standard Error of Mean 2.6
Statistical Analysis 2: Comparison: MPH Discontinuation vs Sustained MPH; Comparison at MPH Maintenance Visit (Week 8); Test type: Superiority; p = .30, t-test, 2 sided; Mean Difference (Final Values) = 2.41, Standard Error of Mean 2.3
Statistical Analysis 3: Comparison: MPH Discontinuation vs Sustained MPH; Comparison at Randomization Phase 1 (Week 9); Test type: Superiority; p = .28, t-test, 2 sided; Mean Difference (Final Values) = 4.01, Standard Error of Mean 3.9
Statistical Analysis 4: Comparison: MPH Discontinuation vs Sustained MPH; Comparison at Randomization Phase 2 (Week 10); Test type: Superiority; p = .00, t-test, 2 sided; Mean Difference (Final Values) = 9.64, Standard Error of Mean 2.5
Statistical Analysis 5: Comparison: MPH Discontinuation vs Sustained MPH; Comparison at Randomization Phase 3 (Week 12); Test type: Superiority; p = .01, t-test, 2 sided; Mean Difference (Final Values) = 7.96, Standard Error of Mean 3.2

2. Primary Outcome: Inhibitory Control Reaction Time Variability (SD of the Reaction Time)
Description: Assessed via the Go/No-Go computerized measure of inhibitory control reaction time variability (with standard deviation of the reaction time being the indicator variability variability). Unit of measure is msec. Minimum is 0, Maximum is 500. Higher scores indicate more variability (higher standard deviation) in reaction time, indicating worse outcome (more characteristic of individuals with ADHD and less characteristic of typically developing individuals).
Time Frame: baseline, study weeks 8, 9, 10 & 12
Population: There was some attrition and missing data at different data collection points.
Measure: Mean (Standard Error); unit: msec
Arm/Group | MPH Discontinuation | Sustained MPH
Number analyzed (Participants) | 85 | 14
msec
  Baseline | 219.6 (17.8) | 196.0 (27.9)
  Maintenance Visit (week 8): number analyzed (Participants) | 72 | 14
  Maintenance Visit (week 8) | 195.9 (17.1) | 199.6 (31.5)
  Randomization 1 (week 9): number analyzed (Participants) | 64 | 13
  Randomization 1 (week 9) | 250.8 (18.8) | 183.8 (37.1)
  Randomization 2 (week 10): number analyzed (Participants) | 59 | 9
  Randomization 2 (week 10) | 288.2 (19.3) | 228.5 (52.8)
  Randomization 3 (week 12): number analyzed (Participants) | 58 | 10
  Randomization 3 (week 12) | 285.2 (20.3) | 199.8 (36.0)
Statistical Analysis 1: Comparison: MPH Discontinuation vs Sustained MPH; Compared at baseline timepoint; Test type: Superiority; p = .32, t-test, 2 sided; Mean Difference (Final Values) = 36.04, Standard Error of Mean 25.4
Statistical Analysis 2: Comparison: MPH Discontinuation vs Sustained MPH; Compared at Maintenance Time Point (week 8); Test type: Superiority; p = .90, t-test, 2 sided; Mean Difference (Final Values) = 4.38, Standard Error of Mean 30.1
Statistical Analysis 3: Comparison: MPH Discontinuation vs Sustained MPH; Compared at Randomization Phase 1 (week 9); Test type: Superiority; p = .007, t-test, 2 sided; Mean Difference (Final Values) = 100.81, Standard Error of Mean 37.5
Statistical Analysis 4: Comparison: MPH Discontinuation vs Sustained MPH; Compared at Randomization Phase 2 (week 10); Test type: Superiority; p = .26, t-test, 2 sided; Mean Difference (Final Values) = 49.07, Standard Error of Mean 56.6
Statistical Analysis 5: Comparison: MPH Discontinuation vs Sustained MPH; Compared at Randomization Phase 3 (week 12); Test type: Superiority; p = .01, t-test, 2 sided; Mean Difference (Final Values) = 123.90, Standard Error of Mean 37.6

3. Primary Outcome: Math Computation - Number of Problems Completed Correctly
Description: Math Computation Curriculum-Based Measure - Number of Problems Completed Correctly. Minimum=0, Maximum=600. Higher scores indicate improved/better performance
Time Frame: baseline, study weeks 8, 9, 10 & 12
Population: There was some attrition and missing data at different data collection points.
Measure: Mean (Standard Deviation); unit: Number of problems completed correctly
Arm/Group | MPH Discontinuation | Sustained MPH
Number analyzed (Participants) | 91 | 17
Number of problems completed correctly
  Baseline: number analyzed (Participants) | 91 | 15
  Baseline | 200.84 (152.8) | 230.93 (127.3)
  Maintenance Visit (week 8): number analyzed (Participants) | 85 | 17
  Maintenance Visit (week 8) | 264.71 (157.4) | 320.12 (142.3)
  Randomization 1 (week 9): number analyzed (Participants) | 81 | 16
  Randomization 1 (week 9) | 221.19 (175.3) | 333.50 (214.1)
  Randomization 2 (week 10): number analyzed (Participants) | 77 | 16
  Randomization 2 (week 10) | 201.69 (164.3) | 323.25 (203.6)
  Randomization 3 (week 12): number analyzed (Participants) | 79 | 16
  Randomization 3 (week 12) | 201.10 (180.3) | 277.51 (190.0)
Statistical Analysis 1: Comparison: MPH Discontinuation vs Sustained MPH; Comparison at Baseline; Test type: Superiority; p = .33, t-test, 2 sided; Mean Difference (Final Values) = 31.13, Standard Error of Mean 32.9
Statistical Analysis 2: Comparison: MPH Discontinuation vs Sustained MPH; Comparison at Maintenance (week 8); Test type: Superiority; p = .06, t-test, 2 sided; Mean Difference (Final Values) = 56.86, Standard Error of Mean 29.5
Statistical Analysis 3: Comparison: MPH Discontinuation vs Sustained MPH; Comparison at Randomization Phase 1 (week 9); Test type: Superiority; p = .05, t-test, 2 sided; Mean Difference (Final Values) = 108.78, Standard Error of Mean 46.8
Statistical Analysis 4: Comparison: MPH Discontinuation vs Sustained MPH; Comparison at Randomization Phase 2 (week 10); Test type: Superiority; p = .008, t-test, 2 sided; Mean Difference (Final Values) = 118.12, Standard Error of Mean 44.2
Statistical Analysis 5: Comparison: MPH Discontinuation vs Sustained MPH; Comparison at Randomization Phase 3 (week 12); Test type: Superiority; p = .07, t-test, 2 sided; Mean Difference (Final Values) = 77.09, Standard Error of Mean 42.9

4. Primary Outcome: % Time on Task
Description: Participants were videotaped while completing the 20-minute Analogue Math task. Their behavior was coded in 20-second intervals by trained coders who determined if the children were on-task or off-task during each interval. The amount of time coded as on-task was divided by the total amount of time and then multiplied by 100 to generate the % of time on task variable.
Time Frame: baseline, study weeks 8, 9, 10, 12
Population: There was some attrition and missing data at different data collection points.
Measure: Mean (Standard Error); unit: percentage of time spent on task
Groups:
- MPH Discontinuation Group: 1. Double-blind (DB) placebo-controlled 4-week methylphenidate (MPH) titration trial. Pts will receive 3 active dosages of MPH (children <25kg: 18mg, 27mg, 36mg; children >25kg: 18mg, 36mg, 54mg for) as well as 1 random week of placebo, given qAM. Pts will begin on the lowest dose (or a randomized placebo week) and proceed through all dose conditions in an incremental fashion.
  2. DB 4-week MPH maintenance phase. The clinician, parent, and teacher ratings of behavior and side effects from the titration trial weeks will be graphed. Two doctors will blindly review the graphs and judge which week was the optimal dose week. Pts will then receive their optimal dose of MPH (qAM) for 4 weeks.
  3. DB 4-week MPH Discontinuation Phase. Pts in this arm will receive placebo (qAM).
  OROS-Methylphenidate (MPH): OROS-methylphenidate will be taken orally once daily at doses that have been approved for the study age group by the U.S. FDA.
- Sustained MPH Group: 1. Double-blind (DB) placebo-controlled 4-week methylphenidate (MPH) titration trial. Pts will receive 3 active dosages of MPH (children <25kg: 18mg, 27mg, 36mg; children >25kg: 18mg, 36mg, 54mg for) as well as 1 random week of placebo, given qAM. Pts will begin on the lowest dose (or a randomized placebo week) and proceed through all dose conditions in an incremental fashion.
  2. DB 4-week MPH maintenance phase. The clinician, parent, and teacher ratings of behavior and side effects from the titration trial weeks will be graphed. Two doctors will blindly review the graphs and judge which week was the optimal dose week. Pts will then receive their optimal dose of MPH (qAM) for 4 weeks.
  3. DB 4-week MPH Discontinuation Phase. Pts in this arm will continue their optimal MPH dose (qAM).
  OROS-Methylphenidate (MPH): OROS-methylphenidate will be taken orally once daily at doses that have been approved for the study age group by the U.S. FDA.
Arm/Group | MPH Discontinuation Group | Sustained MPH Group
Number analyzed (Participants) | 81 | 15
percentage of time spent on task
  Baseline | 74.4 (4.2) | 85.2 (6.4)
  Week 8 (MPH Maintenance dose): number analyzed (Participants) | 79 | 13
  Week 8 (MPH Maintenance dose) | 83.9 (3.8) | 92.7 (3.9)
  Week 9: number analyzed (Participants) | 79 | 14
  Week 9 | 73.1 (3.6) | 91.5 (4.3)
  Week 10: number analyzed (Participants) | 75 | 13
  Week 10 | 69.5 (4.2) | 89.2 (4.2)
  Week 12: number analyzed (Participants) | 76 | 14
  Week 12 | 66.6 (4.5) | 82.6 (6.5)

5. Secondary Outcome: Barkley Sluggish Cognitive Tempo (SCT) Ratings
Description: assessed via parent-completed Barkley Sluggish Cognitive Tempo Scale. Minimum=12, Max=48, higher scores indicate worse outcome.
Time Frame: baseline, study weeks 8, 9, 10 &12
Population: Note: There was some missing data as well as attrition. the numbers of participants with available data for this outcome has been verified.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | MPH Discontinuation | Sustained MPH
Number analyzed (Participants) | 71 | 17
score on a scale
  Baseline (week 1) | 24.41 (1.26) | 24.19 (1.33)
  Maintenance (week 8) | 18.5 (1.1) | 18.2 (1.0)
  Randomization 1 (week 9) | 18.4 (1.2) | 17.5 (1.3)
  Randomization 2 (week 10) | 18.7 (1.1) | 18.0 (1.1)
  Randomization 3 (week 12) | 18.8 (1.1) | 17.6 (1.0)

6. Secondary Outcome: Parent Ratings of Emotional Regulation
Description: assessed via parent-completed Emotion Regulation Checklist (ERC). Outcome assessed is ERC total mean score: minimum value=1, max value=4, higher scores indicate worse outcome
Time Frame: baseline, study weeks 8, 9, 10 &12
Population: There was some attrition and some missing data. # of participants with available data has been verified.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | MPH Discontinuation | Sustained MPH
Number analyzed (Participants) | 71 | 14
score on a scale
  Baseline | 2.1 (0.1) | 2.1 (0.2)
  Maintenance (wk 8) | 1.8 (0.1) | 1.8 (0.1)
  Randomization 1 (wk 9) | 1.8 (0.2) | 1.7 (0.1)
  Randomization 2 (wk 10) | 1.9 (0.1) | 1.8 (0.1)
  Randomization 3 (wk 12) | 1.9 (0.1) | 1.8 (0.1)

7. Secondary Outcome: Spatial Working Memory
Description: Spatial working memory was assessed via the Corsi Computerized Spatial Span Task, which requires the participant to reproduce a sequence of movements by tapping a series of blocks on a computer screen in the same order demonstrated by the examiner. Outcome of interest is total trials correct. Minimum score=0, max score=10. Higher scores indicate better performance.
Time Frame: baseline, study weeks 8, 9, 10 &12
Population: some missing data due to attrition, non-valid trials/responses, and equipment failure. # of participants with available data has been verified.
Measure: Mean (Standard Error); unit: total number of correct trials
Arm/Group | MPH Discontinuation | Sustained MPH
Number analyzed (Participants) | 82 | 16
total number of correct trials
  Baseline | 6.43 (.27) | 6.83 (.33)
  Week 8 (med maintenance) | 6.46 (.25) | 6.63 (.40)
  week 9 | 6.67 (.25) | 7.42 (.42)
  week 10 | 6.54 (.28) | 7.61 (.39)
  week 12 | 6.48 (.29) | 7.24 (.45)

8. Secondary Outcome: Math Reasoning
Description: Math reasoning was assessed by child completion of the AIMSWEB curriculum based measure (CBM) test of Math Concepts and Applications. At baseline (week 1), child's performance was assigned a value of 1.0. The child's performance at weeks 8, 9, 10, and 12 was derived by dividing actual score on the test by the score predicted at that time point after applying the measure's normed "rate of improvement (ROI)" metric to the baseline score. For example, a score of 1.5 at week 8 would indicate that the child's actual score at week 8 was 50% higher than the predicted score at week 8 (which was derived by applying the normed ROI metric to the baseline score). Scores at weeks 8, 9, 10, 12 that are >1.0 indicate greater improvement than expected (so better outcome), while scores at weeks 8, 9, 10, 12 that are <1.0 indicate less improvement than expected (so worse outcome).
Time Frame: baseline, study weeks 1, 8, 9, 10 &12
Population: some missing data due to factors such as attrition and the test not being appropriate to administer all grade levels (e.g., not designed for participants who were in 1st grade) grade. # of participants with available data has been verified.
Measure: Mean (Standard Error); unit: percentage of expected improvement
Arm/Group | MPH Discontinuation | Sustained MPH
Number analyzed (Participants) | 82 | 14
percentage of expected improvement
  Baseline | 1.0 (0.0) | 1.0 (0.0)
  Week 8 | 1.09 (0.06) | 1.27 (0.08)
  week 9 | 1.11 (0.62) | 1.50 (0.15)
  week 10 | 1.15 (0.07) | 1.50 (0.13)
  week 12 | 1.10 (0.06) | 1.65 (0.16)

9. Secondary Outcome: Reading Comprehension
Description: Reading Comprehension was assessed by child completion of the AIMSWEB curriculum based measure (CBM) test of Reading Comprehension. At baseline (week 1), child's performance was assigned a value of 1.0. The child's performance at weeks 8, 9, 10, and 12 was derived by dividing actual score on the test by the score predicted at that time point after applying the measure's normed "rate of improvement (ROI)" metric to the baseline score. For example, a score of 1.5 at week 8 would indicate that the child's actual score at week 8 was 50% higher than the predicted score at week 8 (which was derived by applying the normed ROI metric to the baseline score). Scores at weeks 8, 9, 10, 12 that are >1.0 indicate greater improvement than expected (so better outcome), while scores at weeks 8, 9, 10, 12 that are <1.0 indicate less improvement than expected (so worse outcome).
Time Frame: baseline, study weeks 8, 9, 10 &12
Population: some missing data due to attrition, non-valid test administration. Numbers of participants with available data has been verified.
Measure: Mean (Standard Error); unit: percentage of expected improvement
Arm/Group | MPH Discontinuation | Sustained MPH
Number analyzed (Participants) | 84 | 16
percentage of expected improvement
  baseline | 1.00 (0.0) | 1.00 (0.0)
  week 8 | 1.00 (0.05) | 0.99 (0.11)
  week 9 | 1.02 (0.05) | 1.25 (0.18)
  week 10 | 1.12 (0.05) | 1.27 (0.11)
  week 12 | 1.01 (0.06) | 1.29 (0.14)

10. Secondary Outcome: Written Expression
Description: Assessed by child completion of the AIMSWEB curriculum based measure (CBM) test of Written Expression, with the measure assessing number of words written by the child after receiving a prompt. At baseline (week 1), child's performance was assigned a value of 1.0. The child's performance at weeks 8, 9, 10, and 12 was derived by dividing actual score (# of words written) on the test by the score predicted at that time point after applying the measure's normed "rate of improvement (ROI)" metric to the baseline score. For example, a score of 1.5 at week 8 would indicate that the child's actual score at week 8 was 50% higher than the predicted score at week 8 (which was derived by applying the normed ROI metric to the baseline score). Scores at weeks 8, 9, 10, 12 that are >1.0 indicate greater improvement than expected (so better outcome), while scores at weeks 8, 9, 10, 12 that are <1.0 indicate less improvement than expected (so worse outcome).
Time Frame: baseline, study weeks 1, 8, 9, 10 &12
Population: some missing data due to attrition, non-valid responses, etc. # of participants with available data verified.
Measure: Mean (Standard Error); unit: percentage of expected improvement
Arm/Group | MPH Discontinuation | Sustained MPH
Number analyzed (Participants) | 81 | 17
percentage of expected improvement
  baseline | 1.00 (0.0) | 1.00 (0.0)
  week 8 | 1.16 (0.07) | 0.94 (0.08)
  week 9 | 1.02 (0.07) | 1.06 (0.09)
  week 10 | 1.04 (0.07) | 0.93 (0.08)
  week 12 | 0.91 (0.06) | 1.05 (0.10)

ADVERSE EVENTS:
Time Frame: Duration of trial (3 months)
Description: 1. All-Cause Mortality: The occurrence of death due to any cause.
  2. Serious Adverse Events: adverse events resulting: death, life-threatening event, inpatient hospitalization, significant incapacity, inability to conduct normal functions, or a congenital anomaly. Important medical events may also be considered serious when they require medical or surgical intervention to prevent one of the outcomes listed in this definition.
  3. Other: Adverse events that are not Serious Adverse Events.
Arm/Group | MPH Discontinuation | Sustained MPH
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/92 | 0/17
Other Adverse Events (participants affected / at risk) | 55/92 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPH Discontinuation (N=92) | Sustained MPH (N=17)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) — Participant had suicidal ideation (SI) that the treating psychiatry team deemed related to gender identity issues and bullying and were not judged to be related to study participation. Participant withdrew from study to receive care for SI.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPH Discontinuation (N=92) | Sustained MPH (N=17)
Decreased appetite (Gastrointestinal disorders) | 16 (16) | 10 (10)
Headache (Nervous system disorders) | 6 (6) | 3 (3)
Stomachache (Gastrointestinal disorders) | 8 (8) | 1 (1)
Trouble Sleeping (General disorders) | 13 (13) | 4 (4)
Irritability (Psychiatric disorders) | 17 (17) | 4 (4)
Social Withdrawal (Psychiatric disorders) | 2 (2) | 1 (1)
Sadness (Psychiatric disorders) | 5 (5) | 3 (3)
Dull, tired, listless (General disorders) | 9 (9) | 3 (3)
Skin-picking (Psychiatric disorders) | 13 (13) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Note that the school direct observations outcome was not collected due to data collection not being feasible due to schools' privacy concerns about other students in the classroom. All other outcome measures that were pre-specified Primary or Secondary Outcome Measures have been reported in this ClinicalTrials.gov entry.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT02293655/Prot_SAP_000.pdf